CLINICAL TRIAL: NCT07323693
Title: Clinical Efficacy of Using Bioactive Desensitizer Gel Versus Sodium Fluoride Varnish on Cervical Dentin Hypersensitivity in Adult Patients: A 6m Randomized Clinical Trial
Brief Title: Clinical Efficacy of Using Bioactive Desensitizer Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rawda Hesham Abd ElAziz, Associate Professor, Conservative dentistry department, Faculty of Dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cons 25/4
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Dentin Desensitizing Agents; Dentin Hypersensitivity, Non-carious Cervical Lesions; Dentin Hypersensitivity
Keywords: Dentin hypersentivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioactive Desenstizer (Experimental): A micro-brush applicator was saturated with the material (Predicta Bioactive Desensitizer Gel) and massaged it into the tooth for 30-40 secs.Using a rubbing motion was used to liquefy the gel and allow it to penetrate the surface
  Interventions: Procedure: Treatment
- sodium fluoride varnish (Active Comparator)
  Interventions: Procedure: Treatment

INTERVENTIONS:
Procedure: Treatment — A micro-brush applicator was saturated with the material (Predicta Bioactive Desensitizer Gel) and massaged it into the tooth for 30-40 secs. Using a rubbing motion was used to liquefy the gel and allow it to penetrate the surface
  Arms: Bioactive Desenstizer
Procedure: Treatment — the sodium fluoride (Proshield) varnish, was painted with a disposable micro-brush on the sensitive surface as per the instructions for 60 seconds from the manufacturer.
  Arms: sodium fluoride varnish

SUMMARY:
To evaluate and compare the clinical effectiveness of a Bioactive Desensitizer Gel (which releases calcium and phosphate to form hydroxyapatite) versus a standard 5% Sodium Fluoride (NaF) Varnish in reducing cervical dentin hypersensitivity (CDH) in adult patients over a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* • With ≥1 sensitive tooth and with exposed dentin in the upper or lower dental arches.

  * Grade IV gingival recession.
  * Schiff sensitivity score needed to be ≥2, indicating that application of a jet of air makes the patient respond and move or requests discontinuation of the stimuli application.

Exclusion Criteria:

* • Domestic or in-office fluoride application and bleaching 6 months before beginning of treatment

  * Long-term use of anti-inflammatory, analgesic and psychotropic drugs.
  * Allergies to product ingredients
  * Eating disorders, systemic conditions that cause or predispose patients to develop dentin hypersensitivity (for example, gastroesophageal reflux disease, GERD)
  * Excessive dietary or environmental exposure to acids.
  * Orthodontic appliance treatment within the previous three months.
  * Periodontal surgery within the previous three months before the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | Change from the Baseline, 1 week, 1 months, 3 months, 6 months
  A VAS is a line that is 10 cm in length, the extremes of which represent the limits of pain, a patient may experience an external stimulus (The left endpoint designated no pain was marked as 0 and the right endpoint designated sever pain was marked as 10). Patients will be asked to place a mark on the 10 cm line that indicated their dentin hypersensitivity intensity

SECONDARY OUTCOMES:
Level of Pain Assessment using The Schiff sensitivity scale | Change from the Baseline, 1 week, 1 months, 3 months, 6 months
  It was used to assess dentin hypersensitivity. A score of 0, 1, 2 or 3 was assigned 0 = no subject response to stimulus
  1. = subject response but will continue
  2. = subject responds and moves or requests discontinuation
  3. = painful response to stimulus, discontinuation requested.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No